CLINICAL TRIAL: NCT05517616
Title: A Single-center, Open-label, Single-dose Phase 1 Clinical Study to Investigate the Absorption, Metabolism and Excretion of APG-2575 in Healthy Subjects After Oral Administration of 400 mg/200 µCi [14C] APG-2575 Solution
Brief Title: The Absorption, Metabolism and Excretion of [14C]APG-2575 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG2575XU104
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]APG-2575 (Experimental): To investigate the absorption properties, as well as to evaluate the mass balance and elucidate the pathways of biotransformation after a single oral dose of 400mg, 200μCi [14C] APG-2575 to healthy subjects.
  Interventions: Drug: [14C ]APG-2575

INTERVENTIONS:
Drug: [14C ]APG-2575 — orally, single dose of 400 mg / 200 μCi [14C] APG-2575

SUMMARY:
This study is a single-center, open-label, single-dose clinical pharmacokinetic study. The purpose of this study is to investigate the absorption properties, as well as to evaluate the mass balance and elucidate the pathways of biotransformation after a single oral dose of 400mg, 200μCi [14C] APG-2575 to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-lactating female subjects aged 18-50 (including the boundary value) who have no reproductive needs during the study period and one year after taking the drug;
2. The weight is over 45 kg, and the body mass index (BMI) is between 19 and 26 kg/m2 (including the boundary value);
3. The result of the pregnancy test during the screening period must be negative;
4. The subjects participating in this trial should take effective contraceptive measures with their sexual partners during the study and within 1 year after the end of the research;
5. Subjects must sign the informed consent form voluntarily, agree to abide the requirements of the study protocol.

Exclusion Criteria:

1. After a comprehensive physical examination, vital signs, laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, stool routine, thyroid function), 12-lead electrocardiogram, chest CT, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen and kidney) and other examinations are abnormal and have clinical significance;
2. Resting-corrected QT interval (QTcB) ≥ 450 ms obtained from a twelve-lead electrocardiogram (ECG);
3. Hepatitis B surface antigen or E antigen, hepatitis C virus antibody IgG (Anti-HCV IgG), human immunodeficiency virus antigen/antibody combined test (HIV-Ag/Ab) and Treponema pallidum antibody test positive;
4. The abnormal C-reactive protein of the new coronavirus infection screening has clinical significance or the new coronavirus nucleic acid is positive;
5. Use of any drug that inhibits or induces liver drug metabolizing enzymes within 30 days prior to the screening period
6. Use of any prescription drugs, over-the-counter drugs, herbal medicines, or food supplements, such as vitamins, calcium supplements, within 14 days prior to the screening period;
7. Have any history of clinical serious diseases or diseases or conditions that the investigator considers to be likely to affect the results of the trial , including but not limited to circulatory system, respiratory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic medical history;
8. Reported history or presence of swallowing dysfunction, active gastrointestinal diseases or other diseases that significantly affect drug absorption, distribution, metabolism and excretion;
9. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsades, ventricular tachycardia, atrioventricular block, QT prolongation History of syndrome or symptoms of QT prolongation syndrome and family history (as evidenced by genetic evidence or sudden death of close relatives due to cardiac causes at a young age);
10. Major surgery or surgical incision was not completely healed within 6 months before the screening period; major surgery includes but no limited to any surgery with significant bleeding risk, prolonged general anesthesia, or incisional biopsy or obvious traumatic injury;
11. Allergic constitution, such as those with known history of allergies to two or more substances; or, according to the investigator's judgment, may be sensitive to the investigational drug or its excipients (polyethylene glycol 400, Kolliphor EL, Labrasol, propylene glycol, sodium hydroxide, citric acid;
12. Hemorrhoids or perianal disease with regular/hematochezia, irritable bowel syndrome, inflammatory bowel disease;
13. Habitual constipation or diarrhea;
14. Binge drinking or frequent alcohol consumption within 6 months prior to the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine); or during the screening period Alcohol breath test results > 20 mg/100 mL;
15. Those who smoked more than 5 cigarettes per day or habitually used nicotine-containing products in the first 3 months of the screening period, and were unable to quit during the trial;
16. Drug abuse or use of soft drugs (such as marijuana) 3 months before the screening period or hard drugs (such as cocaine, amphetamines, phencyclidine, etc.) 1 year before the screening period or positive urine drug test during screening period;
17. Those who habitually drink grapefruit juice or excessive tea, coffee and/or caffeinated beverages and cannot quit during the trial;
18. Workers who need to be exposed to radiation for a long time; or have significant radiation exposure (≥2 chest/abdominal CT, or ≥3 other types of X-ray examinations) or participated in clinical trail of radioactivity within 1 year prior to this study.
19. Those with a history of fainting of needles or blood, those with difficulty in blood collection or those who cannot tolerate venipuncture for blood collection;
20. Participated in any other clinical trials (including clinical trials of drugs and devices) within 3 months before the screening period;
21. Those who have been vaccinated within 1 month before screening or who plan to be vaccinated during the study;
22. Those who have lost blood or donated blood up to 400 mL within 3 months before the screening period, or received blood transfusion within 1 month;
23. Subjects with any factors considered inappropriate by the investigator to participate in this trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 6 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration of each blood and plasma sample | Day 1- Day 8
  Use liquid scintillation counter to evaluate Radioactivity concentration of each blood and plasma sample.
Radioactivity concentration in each urine and feces sample. | Day 1- Day 15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each sample.
Number of metabolites and its proportion in plasma, urine and feces. | Day 1- Day 15
  To elucidate the pathways of biotransformation.

SECONDARY OUTCOMES:
Plasma drug concentrations | Day 1- Day 8
  To determine the plasma concentrations of APG-2575 with LC-MS/MS.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Day 1- Day 15
  According to CTCAE v5.0, the number and frequency of adverse events after a single dose of test drug were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China